CLINICAL TRIAL: NCT01913938
Title: Hemophagocytosis in Critically Ill Adult Patients With Cytopenias
Brief Title: Hemophagocytosis in Critically Ill Adult Patients
Acronym: HCIAP
Status: Recruiting | Type: Observational
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Manfred Weiss, Professor, MD, MBA, University of Ulm
Other Study IDs: Hemophagocytosis_Ulm
Record Dates: First submitted 2013-07-29; First posted 2013-08-01 (Estimated); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Hemophagocytosis
Keywords: Hemophagocytosis, adults, rhG-CSF

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, white cells, bone marrow
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with cytopenias: Patients with sepsis and concomitant cytopenias (leukopenia with thrombocytopenia and anemia) who are routinely treated with rhG-CSF will be followed for reconstitution of peripheral blood cell counts. In cooperation with the Department of Hematology, patients are examined for bone marrow cellularity and hemophagocytosis if G-CSF treatment does not result in leukocyte increase.

SUMMARY:
The purpose of the study is to find out whether non-responsiveness to therapeutic recombinant human granulocyte colony-stimulation factor (rhG-CSF) is associated with hemophagocytosis in critically ill adult patients with cytopenias.

DETAILED DESCRIPTION:
In children with bi- or pancytopenia, hemophagocytosis is known as life-threatening hemophagocytic lymphohistiocytosis (HLH). The purpose of the study is to find out whether adult patients with bicytopenia or pancytopenia fulfilling the clinical HLH criteria used in children reflect life-threatening hemophagocytosis and whether hemophagocytosis is associated with responsiveness to recombinant human granulocyte colony-stimulation factor (rhG-CSF) or not.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* critically ill adult patients
* leukopenia and thrombocytopenia
* rhG-CSF therapy

Exclusion Criteria:

* life expectancy < 24 hours
* inclusion in other studies
* trauma patients with reanimation on scene or immediately dying on hospital admission
* pregnancy
* hematologic disorder, malignancy
* high dose corticosteroid treatment or chemotherapy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with leukopenia who are routinely treated with rhG-CSF
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2013-07; Primary Completion 2025-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
responsiveness to recombinant human granulocyte colony-stimulating factor (rhG-CSF) | within 7 days
  increase in leukocytes

SECONDARY OUTCOMES:
8 clinical HLH criteria | 7 days
  degree of fulfillment x out of 8 clinical HLH criteria

OTHER OUTCOMES:
differential blood count, enzymes,biomarkers,immunophenotype | 7 days
  Differential blood count, lactate dehydrogenase, C reactive protein, fibrinogen, triglycerides, ferritin,liver enzymes, aspartate aminotransferase, soluble cluster of differentiation 25, cytokines, procalcitonin biomarkers,immunophenotype (flow cytometry)

CONTACTS AND LOCATIONS:
Overall Officials: Manfred E Weiss, MD, Principal Investigator — Department of Anesthesiology
Locations (2):
- Germany (2):
  - Department of Anaesthesiology, University Hospital Ulm, Ulm
  - Department of Internal Medicine III, Comprehensive Infectious Disease Center, University Hospital Ulm, Germany, Ulm

REFERENCES:
- [Background] Schneider EM, Lorenz I, Muller-Rosenberger M, Steinbach G, Kron M, Janka-Schaub GE. Hemophagocytic lymphohistiocytosis is associated with deficiencies of cellular cytolysis but normal expression of transcripts relevant to killer-cell-induced apoptosis. Blood. 2002 Oct 15;100(8):2891-8. doi: 10.1182/blood-2001-12-0260. PMID 12351400
- [Background] Henter JI, Horne A, Arico M, Egeler RM, Filipovich AH, Imashuku S, Ladisch S, McClain K, Webb D, Winiarski J, Janka G. HLH-2004: Diagnostic and therapeutic guidelines for hemophagocytic lymphohistiocytosis. Pediatr Blood Cancer. 2007 Feb;48(2):124-31. doi: 10.1002/pbc.21039. PMID 16937360
- [Result] Weiss M, Nass M, Schneider EM. Hemophagocytic and/or macrophage activation syndromes may explain thrombocytopenia, leukopenia and anemia in critically ill postoperative/posttraumatic patients. Infection, vol. 39 Suppl. II September, no., pp. S118, 2011.
- [Result] Lorenz MR, Walther P, Weiss M, Huber-Lang M, Schneider EM. Autophagy as a unique biosignature in hemophagocytic cells of patients after major trauma. Infection, vol. 37 (Suppl. III), no. P111, pp. S28 - 29, 2009.
- [Result] Schneider EM, Flacke S, Liu F, Lorenz MR, Schilling P, Nass ME, Foehr KJ, Huber-Lang M, Weiss ME. Autophagy and ATP-induced anti-apoptosis in antigen presenting cells (APC) follows the cytokine storm in patients after major trauma. J Cell Commun Signal. 2011 Jun;5(2):145-56. doi: 10.1007/s12079-010-0113-z. Epub 2011 Jan 13. PMID 21484192
- [Result] Weiss M, Bommer M, Hohmann H, Walther P, Schneider EM. The clinical definition of hemophagocytic lymphohistiocytosis (HLH) as used in children does not explain cytopenia in the majority of critically ill postoperative/posttraumatic patients. Infection 41 Suppl 1: S43 - S44, 2013. DOI 10.1007/s15010-013-0513-0